CLINICAL TRIAL: NCT06446752
Title: A Phase 3 Randomized, Observer-Blind, Placebo-Controlled Study to Assess Efficacy of Meningococcal Group B (rMenB+OMV NZ (Bexsero)) in Preventing Gonococcal Infection Among South African Cis-Gender Women
Brief Title: BIYELA - Bexsero Immunisation in Young Women in Africa
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); University of Witwatersrand, South Africa (Other)
Responsible Party: Principal Investigator, Connie Celum, Professor, Department of Global Health, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: STUDY00019050
Record Dates: First submitted 2024-05-11; First posted 2024-06-06 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-03

CONDITIONS: Gonorrhea; Gonorrhea of Pharynx; Gonorrhea of Anus; Gonorrhea of Cervix
Keywords: sexually transmitted infections; STI; Gonorrhea
MeSH Terms: conditions — Gonorrhea; Sexually Transmitted Diseases | interventions — 4CMenB vaccine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: 1:1 randomization to Bexsero vaccine or placebo injection, to be administered as two intramuscular (IM) doses, two months apart (at Enrollment/Visit 1 and Month 2/Visit 3). Assessment for safety events at one month following the IM doses (Visit 2 and Visit 4), followed by 5 in-clinic follow-up visits for safety, clinical, and laboratory assessments.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind, Placebo-controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Bexsero (Experimental): Meningococcal Serogroup B vaccine rMenB+OMV NZ (Bexsero) administered as an IM injection by 0.5-mL single-dose syringe at enrollment (Visit 1) and 2 months post-enrollment (Visit 3).
  Interventions: Biological: Bexsero
- Placebo (Placebo Comparator): Normal saline (placebo) administered as an IM injection by 0.5-mL single-dose syringe at enrollment (Visit 1) and 2 months post-enrollment (Visit 3).
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Bexsero — Administered as an IM injection by 0.5-mL single-dose syringe at enrollment (Visit 1) and 2 months post-enrollment (Visit 3).
  Other Names: 4MenB-4C
  Arms: Bexsero
Biological: Placebo — Administered as an IM injection by 0.5-mL single-dose syringe at enrollment (Visit 1) and 2 months post-enrollment (Visit 3).
  Other Names: Saline
  Arms: Placebo

SUMMARY:
This proposed 2-arm randomized evaluation of two doses of 4CMenB vaccine versus placebo at Enrollment and Month 2 is designed as a proof-of-concept study to inform potential use for dual meningococcal B and gonococcal prevention, and to inform Neisseria gonorrheae vaccine development.

DETAILED DESCRIPTION:
The World Health Organization (WHO) estimates that the global incidence of gonorrhea in 2020 was 82 million (CI: 48-130 million) among 15 to 49-year-olds, reflecting global incidence rates of 19/1000 women and 23/1000 men in that age group. Most gonococcal infections occur in LMICs. High rates of curable sexually transmitted infections (STIs) have been observed in pre-exposure prophylaxis (PrEP) demonstration projects conducted in adolescent girls and young women (AGYW) from eastern and southern Africa, with prevalences of Chlamydia trachomatis (CT) infection ranging from 24-30%, Neisseria gonorrheae (NG) infection from 7-10%, and syphilis seropositivity from 1-5%.

The consequences of bacterial STIs on AGYW's sexual and reproductive health can be substantial with long-term clinical repercussions: pelvic inflammatory disease (PID), chronic pelvic pain, tubal infertility, pregnancy complications, fetal and neonatal death, and increased susceptibility to HIV. Effective STI prevention interventions are needed to protect individuals, to prevent secondary transmission to partners, and to reduce the risk of long-term reproductive health consequences, particularly for women and their infants. STI prevention interventions could be integrated into PrEP programs, given the high prevalence and incidence of STIs in PrEP populations and the feasibility of providing integrated services in PrEP programs.

N.gonorrhoeae has been identified as a priority pathogen for the development of new vaccines and therapeutics given the current limited therapeutic options in the context of high rates of antimicrobial resistance. A vaccine for NG could mitigate the growing threat of antimicrobial resistance in NG, reduce the high NG prevalence and incidence among African women, and reduce the risk of reproductive morbidity from undiagnosed and untreated NG infection. Women have an increased risk of HIV due to bacterial STIs, both through direct mechanisms such as increased susceptibility due to genital inflammation, and indirectly through infertility, which is associated with increased condom-less sex as part of efforts to become pregnant. There are few other preventative bacterial STI interventions for women on the short-term horizon; unfortunately doxycycline post-exposure prophylaxis for STI prevention (doxy-PEP) was not effective for prevention of CT or NG among 449 Kenyan cis-gender women ages 18 to 30 who were taking HIV PrEP. This lack of efficacy appears to be in part due to adherence; doxycycline was detected in only 29% of 200 hair samples collected at follow-up visits from 50 randomly selected women in the doxy-PEP arm.

Gonorrhea may be vaccine-preventable. Several meningococcal outer membrane vesicle (OMV) proteins have >90% sequence homology with gonococcal OMV proteins. The meningococcal 4CMenB (Bexsero) vaccine (rMenB+OMV NZ), that targets serogroup B N. meningitidis, is a licensed OMV vaccine that contains protein antigens commonly expressed on the surface of both N. meningitidis and N. gonorrhoeae. It induces bactericidal antibodies that mediate killing of the majority of epidemiologically relevant serogroup B N. meningitidis strains. Gonococcal proteins share a high level of identity with several antigens contained in the Bexsero rMenB+OMV NZ vaccine and vaccination with Bexsero induces antibodies in humans that recognize gonococcal proteins 22, 26, 27, 23, 24, 28. In addition to OMV, the vaccine includes three purified recombinant N. meningitidis serogroup B protein antigens (rMenB), two which are fused with accessory antigens: 1) neisserial heparin binding antigen (NHBA), fused with the accessory protein genome-derived neisserial antigen (GNA) 1030, 2) factor H-binding protein (fHbp), fused to GNA2091, and 3) neisserial adhesin A (NadA), presented as a single antigen. NHBA is present in virtually all N. gonorrhoeae strains and its nucleotide and amino acid sequences are highly conserved (96.9% sequence identity in N. gonorrhoeae strains, with 71.3% identity to the Bexsero antigens). Gonococcal fHbp is similar to meningococcal variant 3, which is included in the vaccine, but is not surface exposed and therefore is not expected to contribute to protection. Both GNA2091 and GNA1030 accessory antigens are highly conserved; although their potential contribution to protection is unknown, they could provide an added effect. NadA is absent in gonococcal strains. In a humanized mouse model, 4CMenB immunized mice had antibodies that showed functional activity against NG, clearance of NG was accelerated and bacterial load reduced, serum immunoglobin G (IgG) and IgG cross-reacted with NG OMV and there was a four-fold increase in serum bactericidal50 titres all suggestive of 4CMenB activity against NG28.

ELIGIBILITY:
Inclusion Criteria:

* Individuals born female aged 18-45 years of age inclusive on the day of screening
* In good health as determined by past medical history, medication use, and targeted physical examination,

  1. If not living with HIV, negative HIV test conducted at screening
  2. If living with HIV, on an antiretroviral regimen for ≥3 months, with an undetectable HIV RNA of <200 copies/ml and/or a CD4 count >300 cells/cmm within 12 months of screening
* If of reproductive potential,

  1. Willing to not become pregnant during vaccination period and
  2. Have a negative pregnancy test prior to each vaccination and
  3. Willing to use a reliable method of contraception until month 3 (i.e., after the second vaccination visit)
  4. Not breastfeeding
* Sexually active in the past 3 months, defined as vaginal or anal sex
* At risk for gonorrhea based on sexual behaviour characteristics including

  1. Previous PrEP use in the past 12 months, or
  2. Past history of STIs in the past 12 months, or
  3. 2 or more partners in the past 12 months
* Has provided signed informed consent, and is willing and likely to comply with the trial procedures and follow-up visit requirements
* Has a negative gonorrhea and chlamydia nucleic acid amplification test (NAAT) in the 14 days prior to the Enrollment Visit

Exclusion Criteria:

* Contra-indications to Bexsero
* Previous receipt of a Meningococcal Group B vaccine
* Receipt of antibiotics active against N. gonorrhoeae in the 14 days prior to the Enrollment Visit, including oral or parenteral antibiotics*

  * Participants with NG and/or CT detected at screening may re-screen after receiving appropriate antibiotic treatment
* Planned long-term (> 4 weeks) antibiotic use for prophylaxis or treatment for acne or other bacterial condition(s)
* Use or planned use of a live vaccine within +/- 30 days, an inactive vaccine within +/- 14 days, or an influenza vaccine within +/- 7 days from receipt of study product. Authorized or approved, inactivated COVID-19 vaccines may be given more than 7 days +/- receipt of study product for all study participants
* Use of any investigational drug or vaccine within 30 days prior to enrollment, or planned/anticipated use during study participation
* Currently receiving immunosuppressive agent or systemic corticosteroids (dose >5 mg/day of prednisone) for >14 consecutive days within 90 days prior to enrollment. Topical or inhaled steroids are allowed. Topical steroids cannot be applied to study product injection site
* Has received antineoplastic (chemotherapy) or radiotherapy within 90 days prior to enrollment
* Has received immunoglobulins and/or any blood products within 180 days prior to enrollment
* Progressive, unstable, or uncontrolled disease including but not limited to cardiac, hepatic, renal, immunological, neurological or psychiatric conditions
* Has a condition which in the opinion of the investigator is not suitable for intramuscular vaccination, blood draws, or participation in the trial
* Pregnant or breastfeeding at enrollment

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1100 (Actual)
Dates: Start 2024-08-14 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
First diagnosis of gonorrhea at cervical or anorectal sites occurring greater than or equal to 1 month after the second vaccination with study product through to the study end | 18 months
  Assess efficacy of Bexsero in prevention of cervical and/or anorectal gonococcal infection

SECONDARY OUTCOMES:
First diagnosis of gonorrhea at cervical or anorectal sites occurring >1 month after the second vaccination with study product through to study end, by specified subgroups | 18 months
  To assess efficacy of Bexsero in prevention of cervical and/or anorectal gonococcal infection by pre-specified subgroups, including HIV status, anatomical site (cervical compared to anorectal), and presence or absence of chlamydia
First diagnosis of pharyngeal gonorrhea occurring > 1 month after the second vaccination with study product through to study end, by study arm | 18 months
  To estimate the efficacy of Bexsero in prevention of pharyngeal gonococcal infection
Cumlative GC incidence in the first 9 months after receipt of the second dose of vaccine compared to cumlative GC incidence in the 10-16 months after receipt of the second dose | 18 months
  To assess the durability of protection
To ascertain the safety of Bexsero | 18 months
  Proportion of participants with at least one serious adverse event (SAE), adverse event of special interest (AESI) or other reportable AE (adverse event)

CONTACTS AND LOCATIONS:
Overall Officials: Connie Celum, MD, MPH, Principal Investigator — University of Washington
Locations (5):
- South Africa (5):
  - Desmond Tutu Health Foundation - Emavundleni Research Centre, Cape Town
  - Desmond Tutu Health Foundation - Masiphumulele Site, Cape Town
  - Khayelitsha Vuka Research Clinic, Cape Town
  - Wits RHI Ward 21 Clinical Research Site, Johannesburg
  - Center for Community Based Research (CCBR), Pietermaritzburg

REFERENCES:
- [Background] Celum C, Hosek S, Tsholwana M, Kassim S, Mukaka S, Dye BJ, Pathak S, Mgodi N, Bekker LG, Donnell DJ, Wilson E, Yuha K, Anderson PL, Agyei Y, Noble H, Rose SM, Baeten JM, Fogel JM, Adeyeye A, Wiesner L, Rooney J, Delany-Moretlwe S. PrEP uptake, persistence, adherence, and effect of retrospective drug level feedback on PrEP adherence among young women in southern Africa: Results from HPTN 082, a randomized controlled trial. PLoS Med. 2021 Jun 18;18(6):e1003670. doi: 10.1371/journal.pmed.1003670. eCollection 2021 Jun. PMID 34143779
- [Background] Celum CL, Bukusi EA, Bekker LG, Delany-Moretlwe S, Kidoguchi L, Omollo V, Rousseau E, Travill D, Morton JF, Mogaka F, O'Malley G, Barnabee G, van der Straten A, Donnell D, Parikh UM, Kudrick L, Anderson PL, Haberer JE, Wu L, Heffron R, Johnson R, Morrison S, Baeten JM; POWER Study Team. PrEP use and HIV seroconversion rates in adolescent girls and young women from Kenya and South Africa: the POWER demonstration project. J Int AIDS Soc. 2022 Jul;25(7):e25962. doi: 10.1002/jia2.25962. PMID 35822945
- [Background] Celum CL, Gill K, Morton JF, Stein G, Myers L, Thomas KK, McConnell M, van der Straten A, Baeten JM, Duyver M, Mendel E, Naidoo K, Dallimore J, Wiesner L, Bekker LG. Incentives conditioned on tenofovir levels to support PrEP adherence among young South African women: a randomized trial. J Int AIDS Soc. 2020 Nov;23(11):e25636. doi: 10.1002/jia2.25636. PMID 33247553
- [Background] Kennedy CE, Haberlen SA, Narasimhan M. Integration of sexually transmitted infection (STI) services into HIV care and treatment services for women living with HIV: a systematic review. BMJ Open. 2017 Jun 21;7(6):e015310. doi: 10.1136/bmjopen-2016-015310. PMID 28637733
- [Background] Kakaire O, Byamugisha JK, Tumwesigye NM, Gamzell-Danielsson K. Prevalence and factors associated with sexually transmitted infections among HIV positive women opting for intrauterine contraception. PLoS One. 2015 Apr 10;10(4):e0122400. doi: 10.1371/journal.pone.0122400. eCollection 2015. PMID 25859659
- [Background] Paavonen J, Eggert-Kruse W. Chlamydia trachomatis: impact on human reproduction. Hum Reprod Update. 1999 Sep-Oct;5(5):433-47. doi: 10.1093/humupd/5.5.433. PMID 10582782
- [Background] Ville Y, Leruez M, Glowaczower E, Robertson JN, Ward ME. The role of Chlamydia trachomatis and Neisseria gonorrhoeae in the aetiology of ectopic pregnancy in Gabon. Br J Obstet Gynaecol. 1991 Dec;98(12):1260-6. doi: 10.1111/j.1471-0528.1991.tb15399.x. PMID 1777459
- [Background] Stephens AJ, Aubuchon M, Schust DJ. Antichlamydial antibodies, human fertility, and pregnancy wastage. Infect Dis Obstet Gynecol. 2011;2011:525182. doi: 10.1155/2011/525182. Epub 2011 Sep 22. PMID 21949601
- [Background] Amornkul PN, Vandenhoudt H, Nasokho P, Odhiambo F, Mwaengo D, Hightower A, Buve A, Misore A, Vulule J, Vitek C, Glynn J, Greenberg A, Slutsker L, De Cock KM. HIV prevalence and associated risk factors among individuals aged 13-34 years in Rural Western Kenya. PLoS One. 2009 Jul 31;4(7):e6470. doi: 10.1371/journal.pone.0006470. PMID 19649242
- [Background] Masese L, Baeten JM, Richardson BA, Bukusi E, John-Stewart G, Graham SM, Shafi J, Kiarie J, Overbaugh J, McClelland RS. Changes in the contribution of genital tract infections to HIV acquisition among Kenyan high-risk women from 1993 to 2012. AIDS. 2015 Jun 1;29(9):1077-85. doi: 10.1097/QAD.0000000000000646. PMID 26125141
- [Background] Steen R, Wi TE, Kamali A, Ndowa F. Control of sexually transmitted infections and prevention of HIV transmission: mending a fractured paradigm. Bull World Health Organ. 2009 Nov;87(11):858-65. doi: 10.2471/blt.08.059212. PMID 20072772
- [Background] Naidoo S, Wand H, Abbai NS, Ramjee G. High prevalence and incidence of sexually transmitted infections among women living in Kwazulu-Natal, South Africa. AIDS Res Ther. 2014 Sep 15;11:31. doi: 10.1186/1742-6405-11-31. eCollection 2014. PMID 25243015
- [Background] Ong JJ, Fu H, Baggaley RC, Wi TE, Tucker JD, Smith MK, Rafael S, Falconer J, Terris-Prestholt F, Mameletzis I, Mayaud P. Missed opportunities for sexually transmitted infections testing for HIV pre-exposure prophylaxis users: a systematic review. J Int AIDS Soc. 2021 Feb;24(2):e25673. doi: 10.1002/jia2.25673. PMID 33605081
- [Background] Ong JJ, Baggaley RC, Wi TE, Tucker JD, Fu H, Smith MK, Rafael S, Anglade V, Falconer J, Ofori-Asenso R, Terris-Prestholt F, Hodges-Mameletzis I, Mayaud P. Global Epidemiologic Characteristics of Sexually Transmitted Infections Among Individuals Using Preexposure Prophylaxis for the Prevention of HIV Infection: A Systematic Review and Meta-analysis. JAMA Netw Open. 2019 Dec 2;2(12):e1917134. doi: 10.1001/jamanetworkopen.2019.17134. PMID 31825501
- [Background] Tacconelli E, Carrara E, Savoldi A, Harbarth S, Mendelson M, Monnet DL, Pulcini C, Kahlmeter G, Kluytmans J, Carmeli Y, Ouellette M, Outterson K, Patel J, Cavaleri M, Cox EM, Houchens CR, Grayson ML, Hansen P, Singh N, Theuretzbacher U, Magrini N; WHO Pathogens Priority List Working Group. Discovery, research, and development of new antibiotics: the WHO priority list of antibiotic-resistant bacteria and tuberculosis. Lancet Infect Dis. 2018 Mar;18(3):318-327. doi: 10.1016/S1473-3099(17)30753-3. Epub 2017 Dec 21. PMID 29276051
- [Background] Stewart J, Bukusi E, Sesay FA, Oware K, Donnell D, Soge OO, Celum C, Odoyo J, Kwena ZA, Scoville CW, Violette LR, Morrison S, Simoni J, McClelland RS, Barnabas R, Gandhi M, Baeten JM. Doxycycline post-exposure prophylaxis for prevention of sexually transmitted infections among Kenyan women using HIV pre-exposure prophylaxis: study protocol for an open-label randomized trial. Trials. 2022 Jun 16;23(1):495. doi: 10.1186/s13063-022-06458-8. PMID 35710444
- [Background] Petousis-Harris H, Radcliff FJ. Exploitation of Neisseria meningitidis Group B OMV Vaccines Against N. gonorrhoeae to Inform the Development and Deployment of Effective Gonorrhea Vaccines. Front Immunol. 2019 Apr 9;10:683. doi: 10.3389/fimmu.2019.00683. eCollection 2019. PMID 31024540
- [Background] Semchenko EA, Tan A, Borrow R, Seib KL. The Serogroup B Meningococcal Vaccine Bexsero Elicits Antibodies to Neisseria gonorrhoeae. Clin Infect Dis. 2019 Sep 13;69(7):1101-1111. doi: 10.1093/cid/ciy1061. PMID 30551148
- [Background] Hadad R, Jacobsson S, Pizza M, Rappuoli R, Fredlund H, Olcen P, Unemo M. Novel meningococcal 4CMenB vaccine antigens - prevalence and polymorphisms of the encoding genes in Neisseria gonorrhoeae. APMIS. 2012 Sep;120(9):750-60. doi: 10.1111/j.1600-0463.2012.02903.x. Epub 2012 Apr 28. PMID 22882265
- See also: Global progress report on HIV, viral hepatitis and sexually transmitted infections, 2021 — https://iris.who.int/bitstream/handle/10665/342808/9789240030985-eng.pdf